CLINICAL TRIAL: NCT03137342
Title: Pepped on Pre-exposure Prophylaxis (PrEP): Pilot-randomized Controlled Trial (RCT) to Assess the Feasibility/Acceptability of the Pepped-for-PrEP Package (Counseling and Problem-solving PrEP Adherence Intervention With Behavioral Activation (BA) Approach) Among Stimulant Abusing MSM.
Brief Title: Pepped on Pre-exposure Prophylaxis (PrEP): A Counseling and Problem-Solving PrEP Adherence Intervention for Stimulant Using Men Who Have Sex With Men (MSM).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, Professor, Departments of Behavioral & Social Health Sciences and Epidemiology, School of Public Health Professor, Department of Psychiatry & Human Behavior, Alpert Medical School Director, Center for Health Equity Research (CHER), Brown University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 1610001629
Record Dates: First submitted 2017-04-04; First posted 2017-05-02 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: PrEP Uptake; Stimulant Abuse; Adherence, Medication
Keywords: PrEP; Adherence; Risk Reduction; Stimulant Use
MeSH Terms: conditions — Medication Adherence; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Intervention Condition: Pepped-for-PrEP intervention counseling plus standard of care adherence counseling as part of their PrEP related care via The Miriam Hospital Control Condition: only the standard of care adherence counseling as part of their PrEP related care via The Miriam Hospital.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blind to the participant's assigned intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pepped on PrEP (Experimental): Using an efficient stepped care ("adaptive") model, all participants will receive three sessions of PrEP-STEPS counseling for PrEP adherence delivered by a Masters-level or above therapist. Some individuals may require a more intensive approach. These participants will receive an additional seven counseling sessions of behavioral activation with integrated cognitive behavioral therapy (CBT) designed to reduce stimulant use and promote positive behaviors.
  Interventions: Behavioral: Pepped on PrEP Package
- Standard of Care (No Intervention): PrEP adherence counseling from the Miriam Hospital PrEP Clinic.

INTERVENTIONS:
Behavioral: Pepped on PrEP Package — A counseling and problem-solving adherence intervention with a Behavioral Activation approach to re-engage participants in safe but pleasurable activities in life and addresses stimulant abuse as well as associated factors, including depression, as barriers to optimal PrEP adherence.
  Arms: Pepped on PrEP

SUMMARY:
Pepped on PrEP is an innovative pilot RCT designed by an interdisciplinary team to develop a counseling and problem-solving PrEP adherence intervention with a Behavioral Activation (BA) approach that aims to re-engage participants in safe but pleasurable activities in life and addresses stimulant-abuse as well as associated factors including depression, as barriers to optimal PrEP adherence.

DETAILED DESCRIPTION:
Enrolled participants will receive a referral to the Miriam Hospital for standard of care PrEP treatment. Once prescribed PrEP through the Miriam Hospital, the study participants will be randomly assigned to one of two treatment conditions. In the intervention condition, participants will receive a two-stepped intervention which could include up to 10 free BA and risk reduction (RR) counseling sessions. Participants assigned to the comparison condition will receive the standard of care for PrEP treatment at the Miriam Hospital, which includes information about PrEP and how to obtain it, assistance from medical staff in obtaining health insurance for study participants, and information regarding local community resources.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or older
2. Sex: assigned male sex at birth
3. Self-reports having sex with another man in the past month while using stimulants
4. Self-reports behavioral risk for HIV infection (consistent with the Center for Disease Control guidelines) for prescribing PrEP: condomless anal intercourse with at least one HIV-infected or unknown serostatus partner in the preceding six months)
5. Not currently prescribed PrEP at initial visit
6. Able to speak and understand English (for consenting and counseling)
7. Lives in New England

Exclusion Criteria:

1.) Potential participants unable to provide informed consent, including people with severe mental illness requiring immediate treatment or with mental illness limiting their ability to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men and report stimulant use at screening
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
PrEP Uptake | Baseline Stage 2
  >80% of participants who complete Stage 1 baseline and report PrEP initiation (verified by prescription) will progress to Stage 2 Baseline.
Improve rate of PrEP adherence | Daily beginning at Stage 2 Baseline up to the four month assessment visit
  Wisepill electronic pill dispenser will monitor when the pill dispenser is opened to measure medication adherence .
Improve rate of PrEP adherence | Baseline Stage 2 and four month assessment
  Self report adherence to assess for change in adherence.

SECONDARY OUTCOMES:
Reduce Unsafe Sex | Baseline Stage 1,Baseline Stage 2 and four month assessment
  Self report sexual history to assess for change in sexual risk.
Reduce Stimulant Use | Baseline Stage 1,Baseline Stage 2 and four month assessment
  Self report stimulant use to assess for change in drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Mimiaga, ScD, MPH, Principal Investigator — Brown University, School of Public Health, Center for Health Equity Research
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes